CLINICAL TRIAL: NCT04868552
Title: The Effect of Universal Pre-hospital Naloxone Education on Patient and Family Safety, Attitudes and Experience in the Surgical Patient: a Prospective Randomized Trial
Brief Title: Naloxone Education in Total Joint Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-19-474
Record Dates: First submitted 2019-10-07; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Opioid Use; Pain, Musculoskeletal; Surgery; Overdose of Opiate
Keywords: naloxone; patient education; joint arthroplasty
MeSH Terms: conditions — Musculoskeletal Pain; Opiate Overdose

STUDY DESIGN:
Intervention Model Description: prospective randomized
Who Masked: Outcomes Assessor
Masking Description: investigators analyzing data will not know whether participants are in the intervention or no-intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naloxone education (Experimental): These participants will receive a pre-hospital naloxone education module during their pre-operative joint class
  Interventions: Other: Pre-hospital naloxone education
- Standard Education (No Intervention): These participants will receive the standard pre-hospital education including pain management and opioid safety, but will not specifically be given the new naloxone-education module in the pre-hospital setting

INTERVENTIONS:
Other: Pre-hospital naloxone education — a 5-10 minute pre-hospital education module teaching patients and support persons how and when to administer naloxone
  Arms: Naloxone education

SUMMARY:
This study examines the efficacy of a brief pre-hospital naloxone education module added to the standard "Total Joint Class" curriculum on patient safety and experience. Participants will consist of 250 patient-and-support-person pairs. The primary outcome is "readiness to use" naloxone - a proxy for opioid overdose safety. Patient factors contributing to this primary outcome as well as the effect on patient attitude and experience will also be investigated.

DETAILED DESCRIPTION:
Opioids are powerful pain medications which currently serve a necessary role in recovery after knee or hip replacement surgery. However, opioids also pose a danger to both the patient and to other members of the household in the event of accidental overdose because they can cause respiratory depression and death. To minimize the risk of opioid overdose, patients are educated in appropriate use and storage of their medication. They are also provided with a prescription for naloxone. Naloxone is an emergency-use, potentially life-saving antidote to opioid pain medication. It can be sprayed into the nostrils of the opioid overdose victim by a non-medically trained bystander while waiting for the ambulance to arrive, and can make the difference between life and death for a child or adult. However, only about 30% of patients choose to fill their naloxone prescription when they go home from hospital after joint replacement surgery at Carilion Roanoke Memorial Hospital. The first purpose of this study is to evaluate whether teaching patients about opioid overdose and naloxone treatment influences whether patients fill their naloxone prescription and whether they can appropriately administer naloxone in the event of an overdose in the home. Additionally, this study will look at what factors, other than pre-surgery education, influence whether a patient fills their naloxone prescription or not. The resources available for opioid overdose prevention in the community are limited, and this study will help guide the effective use of those resources.

The participants in this study will be patients who are planning hip or knee replacement surgery. They will enroll together with their primary support person. Two hundred and fifty patient and primary-support-person pairs will be enrolled prospectively over a 9-month period. All participant pairs will be randomized to receive either only the current three-hour pre-operative Joint Class (which is mandatory for all patients with their support person and includes education on opioids and pain management), or to receive, in addition, a new educational module. The new module will consist of a modified version of the REVIVE! Course, a course designed for people without prior medical training on the recognition of an opioid overdose and appropriate response including naloxone administration. Participants will be asked to complete an enrollment questionnaire prior to the educational intervention, a 2-week Recovery Journal (pain and medication diary) following surgery, and a follow-up questionnaire at the first post-operative visit, 2 weeks after surgery. Patients will also receive a short, 3-4 item questionnaire 6 months after surgery to collect data on the risk of long-term opioid use and the outcome of the naloxone in the home.

Demographic and clinical data that is collected will be used to describe the study population and determine factors that act as barriers to effective opioid overdose reversal with naloxone in the home. This study will also examine the influence of education on the experience of the patient within the healthcare system, attitudes of patients towards opioids and naloxone, and patient safety. Standardized assessments that will be used to address these study questions include the Opioid Overdose Knowledge Scale (OOKS), the Opioid Overdose Attitude Scale (OOAS), and the PROMIS Pain Medication Misuse, Pain Intensity, and Pain Interference short forms.

There are few studies that examine the influence of naloxone education for the layperson, so evidence in this field is limited. This study is unique in that it moves the conversation from the arena of chronic pain management and opioid addiction and focuses on the population of patients managing acute pain before and after surgical procedures. Outcomes of this research will help to direct prevention resources by answering very topical questions about the usefulness and effects of naloxone co-prescription with opioids for acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients and "primary support person" pairs in which
* the patient is planning total or partial elective hip replacement at Carilion Roanoke Memorial Hospital OR
* the patient is planning total or partial elective knee replacement at Carilion Roanoke Memorial Hospital OR
* willingness to participate in study activities

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Poor cognitive function
* Poor English language skills
* Inmate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
"Readiness to Use Naloxone" assessed by survey and Opioid Overdose Knowledge Scale administration | approximately 2 weeks (from surgery to first follow-up visit)
  This measure is expressed as a binary yes/no for each patient-support person pair. It can be assessed with the survey tool used at the patient's follow up appointment. The patient/ support person pair must satisfy each of the three following conditions.
  1. patient reports naloxone is present in the home (or carried with the patient) (assessed by Y/N question)
  2. the support person reports knowledge of and immediate access to the naloxone (assessed by Y/N question)
  3. the support person demonstrates competency for naloxone administration by scoring a passing mark on the modified Opioid Overdose Knowledge Scale (OOKS) (Williams et al. 2013). For our purposes, this will be a score greater than or equal to 34/45.
  If the three conditions are met, then the pair is assessed a "yes" score on "Readiness to Use Naloxone". If any condition is not met, then the pair is assessed a "no" score on "Readiness to Use Naloxone".

SECONDARY OUTCOMES:
Correlation between indication for surgery (described by International Classification of Diseases 9/10 code) and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  "Readiness to Use Naloxone" as described in our primary outcome measure will be used in the majority of our secondary outcomes. It functions as a binary variable.
  Indications for surgery are described by International Classification of Diseases 9/10, which are categorical variables with a uniform unit of measure. These codes are entered into the patient's electronic medical record by the patient's surgeon and would be retrieved by a study team member. Codes expected to be present in the study include:
  Musculoskeletal 16-Osteoarthritis of the Hip Musculoskeletal 17-Osteoarthritis of the Knee
Correlation between procedure (Current Procedural Terminology code) and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  "Readiness to Use Naloxone" as described in our primary outcome measure will be used in the majority of our secondary outcomes. It functions as a binary variable.
  The operations that patients undergo are described by Current Procedural Terminology codes, which are categorical variables with a uniform unit of measure. These codes are entered into the patient's electronic medical record by the patient's surgeon and would be retrieved by a study team member. Codes expected to be present in the study include:
  1005073- Arthroplasty, knee, condyle and plateau 27130 - Arthroplasty, acetabular and proximal femoral prosthetic replacement (total hip arthroplasty), with or without autograft or allograft
Correlation between patient comorbidities (described by International Classification of Diseases 9/10 code and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  "Readiness to Use Naloxone" as described in our primary outcome measure will be used in the majority of our secondary outcomes. It functions as a binary variable.
  Comorbidities are other elements of a patient's health that are identified by their primary care physicians or other specialists. These comorbidities International Classification of Diseases 9/10, which are categorical variables with a uniform unit of measure. These codes are entered into the patient's electronic medical record by the patient's surgeon and would be retrieved by a study team member. Codes expected to be present in the study include:
  Musculoskeletal 16-Osteoarthritis of the Hip Musculoskeletal 17-Osteoarthritis of the Knee
correlation between patient age and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  age (exploratory analysis)
correlation between patient sex and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  sex (exploratory analysis)
correlation between patient race and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  race (exploratory analysis)
correlation between patient ethnicity and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  ethnicity (exploratory analysis)
correlation between patient household income and "Readiness to Use Naloxone" | 2 months (time from study enrollment to first post-op visit)
  household income (exploratory analysis)
Amount of opioid used at home | 7 months (time from enrollment to 6 month follow-up phone call)
  milligrams of morphine equivalents
Post-operative pain as measured by the Patient Reported Outcome Measurement Information System Pain Interference 6a assessments | 7 months (time from enrollment to 6 month follow-up phone call)
  Each question usually has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For the adult 6-item form, the lowest possible raw score is 6; the highest possible raw score is 30 (see all short form scoring tables in Appendix 1). All questions must be answered in order to produce a valid score using the scoring tables. If a participant has skipped a question, use the HealthMeasures Scoring Service (https://www.assessmentcenter.net/ac_scoringservice) to generate a final score. Locate the applicable score conversion table in Appendix 1 and use this table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Post-operative pain as measured by the Patient Reported Outcome Measurement Information System Pain Intensity 3a | 7 months (time from enrollment to 6 month follow-up phone call)
  Each question has five response options ranging in value from one to five. To find the total raw score for the short form, sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15.
  For most Patient-Reported Outcomes Measurement Information System instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. The T-score is provided with an error term (Standard Error or SE). The Standard Error is a statistical measure of variance and represents the "margin of error" for the T-score.
  Important: A higher Patient-Reported Outcomes Measurement Information System T-score represents more of the concept being measured.
High risk behavior as measured by the Patient Reported Outcome Measurement Information System Pain Medication Misuse assessment | 7 months (time from enrollment to 6 month follow-up phone call)
  Each question has five response options ranging in value from one to five. To find the total raw score for the short form, sum the values of the response to each question. For this instrument, the lowest possible raw score is 7; the highest possible raw score is 35. All questions must be answered in order to produce a valid score.
  For most Patient-Reported Outcomes Measurement Information System instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. The T-score is provided with an error term (Standard Error or SE). The Standard Error is a statistical measure of variance and represents the "margin of error" for the T-score.
Patient and caregiver knowledge | 7 months (time from enrollment to 6 month follow-up phone call)
  Opioid Overdose Knowledge Scale: The Opioid Overdose Knowledge Scale items use a 'yes/no or don't know'; or 'true/false or don't know' response format.
  Each correct answer scores one point. 'Don't know' and incorrectly marked responses (mistakes) are scored zero. Total score range: 0-45 points.
  OPIOID OVERDOSE KNOWLEDGE SCALE (OOKS):
  INSTRUCTIONS
  Total Score (45 items):
  One point if marked (33 Correct/True items): 1a, 1b, 1c, 1d, 1e, 1f, 1g, 1h, 1i, 2b, 2c, 2d, 2e, 2g, 2h, 3a, 3b, 3d, 3f, 3g, 3i, 3j, 4a, 5a, 5b, 5c, 6a, 7a, 8b, 9T, 11T, 12T, 14T One point if NOT marked (12 Incorrect/False items): 2a, 2f, 2i, 2j, 3c, 3e, 3h, 3k, 5d, 5e, 10F, 13F. You might chose to use the 'record into same variables' function of Statistical Package for the Social Sciences and inverse the values of these items.
Patient and caregiver attitude | 7 months (time from enrollment to 6 month follow-up phone call)
  Opioid Overdose Attitude Scale: SCORING The Opioid Overdose Attitude Scale is scored continuously using a 5-point Likert scale: completely disagree (1 point), disagree (2 points), unsure (3 points), agree (4 points) and completely agree (5 points).
  Reverse negative items:
  The following negative items need to be reversed before computing the total of scale points: 4, 6, 7, 9, 11, 15, 16, 17, 18, 23, 24, 25. You can use the 'record into same variables'
  OPIOID OVERDOSE ATTITUDES SCALE (OOAS):
  INSTRUCTIONS function of Statistical Package for the Social Sciences. Recode these items as: completely disagree (5 point), disagree (4 points), unsure (3 points), agree (2 points) and completely agree (1 points).
  Totals Scores:
  Once negative items have been reversed, add all items' points. The total scale points can range from 28 to 140 points.
Prescription fill rate | approximately 2 weeks (from surgery to first follow-up visit)
  patient reports naloxone is present in the home (or carried with the patient)
Naloxone accessibility | approximately 2 weeks (from surgery to first follow-up visit)
  "yes/no" answer to the question: "Do you know where naloxone is stored in the home and have immediate access to it in an emergency?"
Rescuer competence measured by modified Opioid Overdose Knowledge Scale Score (see outcome 14 for scoring) | approximately 2 weeks (from surgery to first follow-up visit)
  the support person demonstrates competency for naloxone administration by scoring a passing mark (34/45) on the modified Opioid Overdose Knowledge Scale

CONTACTS AND LOCATIONS:
Overall Officials: Cassandra Mierisch, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Institute for Orthopedics and Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No